CLINICAL TRIAL: NCT00836316
Title: Effects of Intraperitoneal Levobupivacaine on Pain After Laparoscopic Cholecystectomy: A Prospective, Randomized, Double-Blinded Study
Brief Title: Levobupivacaine During Cholecystectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ege University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LDC-2008
Record Dates: First submitted 2009-02-03; First posted 2009-02-04 (Estimated); Last update posted 2009-02-04 (Estimated); Status verified 2009-02

CONDITIONS: Cholelithiasis; Pain
Keywords: laparoscopic cholecystectomy
MeSH Terms: conditions — Cholelithiasis; Pain | interventions — Levobupivacaine

INTERVENTIONS:
Drug: levobupivacaine — intraperitoneal administration of levobupivacaine on pain after laparoscopic cholecystectomy

SUMMARY:
The purpose of this study is to determine the effects of intraperitoneal administration of levobupivacaine on pain after laparoscopic cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:

* cholelithiasis
* chronic cholecystitis

Exclusion Criteria:

* hypersensitivity to local anesthetics
* acute cholecystitis
* morbid obesity

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University School of Medicine, Izmir, Turkey (Türkiye)